CLINICAL TRIAL: NCT00350649
Title: Maximizing the Efficacy of Cognitive Behavior Therapy and Contingency Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0407026913
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Marijuana Dependence
Keywords: behavior modification; cognitive behavioral therapy; combination therapy; drug abuse therapy; drug addition; human therapy evaluation; psychotherapy; clinical trial phase II; coping; drug and alcohol abstinence; longitudinal human study; outcomes research; outpatient care; psychological reinforcement; therapy compliance; behavior and social research tag; human subjects; neuropsychological test; patient oriented research
MeSH Terms: conditions — Marijuana Abuse; Alcohol Abstinence; Patient Compliance; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): manualized delivery of CBT by trained clinicians
  Interventions: Behavioral: Standard CBT
- 2 (Active Comparator): CBT with Contingency Management reinforcement for attendance and completing homework (CBT+CM/adherence)
  Interventions: Behavioral: CBT+CM/adherence
- 3 (Experimental): Contingency Management for abstinence alone (CM/abstinence)
  Interventions: Behavioral: CM/abstinence
- 4 (Active Comparator): Contingency Management integrated with CBT (CM/abstinence+CBT)
  Interventions: Behavioral: CM/abstinence+CBT

INTERVENTIONS:
Behavioral: Standard CBT — Manualized delivery of CBT by trained clinicians
  Arms: 1
Behavioral: CBT+CM/adherence — CBT and Clinical Management for attendance and completing homework
  Arms: 2
Behavioral: CM/abstinence — Contingency Management
  Arms: 3
Behavioral: CM/abstinence+CBT — Contingency Management for abstinence in addition to manualized CBT delivered by a trained clinician
  Arms: 4

SUMMARY:
Cognitive-behavioral coping skills therapy (CBT) is a widely used and recognized treatment that has been empirically validated for a range of substance use disorders, often with emergent effects and continuing improvement even after treatment ends. Treatment retention and compliance are associated with enhanced treatment outcomes in CBT. Contingency management (CM) also has very strong support and is associated with rapid, robust effects on targeted outcomes. Despite their many strengths, neither CBT nor CM is universally effective. It is now essential to seek strategies to maximize and extend the effectiveness of these two approaches and to better understand how these treatments exert their effects.

DETAILED DESCRIPTION:
The investigators propose to evaluate targeted strategies to maximize the effectiveness of CBT and CM, respectively. To maximize the effectiveness of CBT, the investigators will evaluate the benefit of adding CM, with reinforcement for session attendance and homework completion, to standard individual CBT for outpatient marijuana abusers, in order to expose participants to more skill training and opportunities for practice of skills. To maximize the effectiveness and durability of CM, we will evaluate the benefit of integrating it with skills training, specifically designed to reduce drop off effects, in order to extend CM's benefits beyond the active treatment period. We propose to conduct a Stage II trial which will: (1) Evaluate the efficacy of four conditions for 160 marijuana dependent outpatients: (a) Standard CBT, (b) CBT with CM reinforcement for attendance and completing homework (CBT+CM/adherence), (c) CM for abstinence alone (CM/abstinence), (d) CM for abstinence integrated with CBT (CM/abstinence+CBT), and (2) Evaluate the longer-term durability and / or delayed emergence of treatment effects after termination of the study treatments through a one-year follow-up. Secondary aims will be to conduct (a) detailed process studies to evaluate whether the proposed enhancements affect proximal and distal outcomes as hypothesized and (b) economic analyses. Study treatments will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 year old marijuana dependent
* willing to sign consent
* no use of prescribed psychotropic drugs
* willing to give three individuals as contacts
* willing to accept randomization
* read and write English (third grade level)

Exclusion Criteria:

* unable to commit to 1 year follow up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2004-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Self reported marijuana use (days of abstinence by week) and results of urine toxicology screens | 12 weeks

SECONDARY OUTCOMES:
Economic analysis with use of PACC-SAT | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Carroll, PhD, Principal Investigator — Yale University
Locations (1):
- ASAP/1 Long Wharf, New Haven, Connecticut, United States